CLINICAL TRIAL: NCT06557382
Title: The Power of Cognitive Skills to Predict Reading Speed
Brief Title: Cognitive Skills and Reading Speed
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ozden erkan, assistant professor, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-8008
Record Dates: First submitted 2024-08-09; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Function 1, Social; Reading Problem
Keywords: cognitive skills; predict reading speed; child
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary school 1st grade students: Cognitive tests and reading-related evaluations will be administered to illiterate first-grade primary school students before and 6 months after they start education.
  Interventions: Behavioral: Cognitive tests and reading-related evaluations

INTERVENTIONS:
Behavioral: Cognitive tests and reading-related evaluations — Tests assessing cognitive status and reading were administered. (Frankfurter; MVPT-3, TILLs; etc.)

SUMMARY:
The aim of this study is to examine the relationship between cognitive skills, reading speed and reading comprehension skills in children who will learn to read and who do not have any diagnosis.

DETAILED DESCRIPTION:
Learning to read is a very difficult process for both parents and children. Some children overcome this process more easily, while others have more difficulty. Understanding this process and the factors that affect it is important for developing academic skills. Reading is a complex, multifactorial, and dynamic process. When reading begins, parallel activation of limbic, motor, and cognitive processes occurs in different brain regions, including the cortex, thalamus, and basal ganglia. Orthographic word processes, phonological analysis, mapping between print, sound, and meaning, articulatory registration, and semantic/syntactic processing of written words occur through activation of left ventral occipitotemporal, dorsal temporoparietal, and left inferior frontal brain networks. During this process, the brain mentioned above networks establish connections with many areas of both hemispheres to enable comprehension. Reading skills involve the activation and interaction of cognitive processes such as attention, working memory, and executive control. Their study with 9-year-old children stated that planning skills are important for reading and that good inhibitory control increases phonotic coding skills. Miller and colleagues noted that the executive function subcomponents of working memory, but not inhibition, explained 52% of the variance in literacy and 81% of the variance in mathematics. Gallen and colleagues found that the ability to sustain attention was associated with reading and mathematics skills. McClelland and colleagues suggested that children with a higher standard deviation score in attention span at age 4 were 48.7% more likely to graduate from college by age 25. As can be seen, although reading skills have been linked to cognitive abilities in the literature, complete clarity has not been achieved. It would be appropriate to evaluate reading in general as word recognition/identification and reading comprehension skills. While word recognition involves lower-level cognitive processes, comprehension requires the automatization of lower-level cognitive skills coordinated with the effect of higher-level cognitive skills. In this context, it may be necessary to examine which cognitive skill can predict reading according to subheadings of reading such as reading speed and reading comprehension. If the relationship between cognitive skills and the speed of learning to read and reading comprehension is revealed, the performance of children at risk of falling behind in reading can be increased with additional measures. Since it will be predicted which of the children who have just started school will fall behind in learning to read by using the tests with high prediction coefficients to be determined at the end of the study, developmental measures can be taken for these children. In addition, it will be possible to focus on cognitive exercises to increase the success of these children in their educational lives.

The purpose of this study is to examine the relationship between cognitive skills in children who will learn to read and who do not have any diagnosis and reading speed and reading comprehension skills.

ELIGIBILITY:
Inclusion Criteria:

* Being 6 years old and above and starting primary school
* Not knowing how to read and write
* Not having received any previous literacy training
* Knowing Turkish

Exclusion criteria:

* Having dyslexia
* Being diagnosed with a neurological or psychiatric disease
* Having an organic disorder such as hearing and vision

Ages: 72 Months to 96 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — ALL GENDER
Study Population: Primary School Students Aged 6-8.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Frankfurter tests | Baseline and 6 months after initial evaluation
  The reliability and validity studies of the Frankfurter Concentration Test for five-year-old children, developed by Raatz and Möhling (1971). were conducted in Germany.It is a short, simple test that measures attention and concentration skills. It is a performance test that involves marking a target stimulus in a visual.
Cancellation Test | Baseline and 6 months after initial evaluation
  It is a neuropsychological test developed by Weintraub and Mesulam (1985). The IT in the BILNOT Battery has been standardized for both adults and children. In studies conducted in our country, it has been observed that the IT scores are grouped under the factors of visual-spatial scanning, impulsivity and reaction speed regarding the stimulus context.
Executive Functions and Occupational Routines Scale (EFORTS) | Baseline and 6 months after initial evaluation
  It evaluates the mental characteristics of children aged 6-12, such as impulse, verbal and non-verbal memory, self-regulation, problem solving, and planning. It is scored by the family on a 1-5 Likert scale. It has 3 subsections, including morning-evening routines, play-fun, and social routines, and contains a total of 30 questions.
Forward and Backward Digit Span | Baseline and 6 months after initial evaluation
  To assess working memory, the Digit Span Subtest of the Wechsler Intelligence Scale for children was used ın forward digit span, the child is told a 2-digit number and asked to repeat it. When the same digit is repeated twice correctly, the number of digits is increased. The number of digits is increased until an error is made. When an error is made twice, the test is finished and the forward digit span is determined. The backward digit span is similar to the forward digit span. The only difference is that the child is asked to repeat the given numbers backwards.
The Head-Toes-Knees-Shoulders | Baseline and 6 months after initial evaluation
  It measures children's ability to regulate their behavior. Children are asked to do the opposite of what is said. The task increases in complexity by including 4 body parts (head, toe, knee and shoulder). Answers are scored from 0 to 2 points.
Motor-free Perception Test (MVPT-3). | Baseline and 6 months after initial evaluation
  MVPT-3 includes all visual perception subheadings. The test consists of 9 subfields and 65 shapes, namely visual discrimination (1-8), shape formation (9-13), visual memory-I (14-21), visual proximity-I(22-34), visual discrimination (35-45), position in space (46-50), figure-ground (51-55), visual proximity-II (56-60) and visual memory-II (61-65). Total visual perception score is calculated.
Test of Integrated Language and Literacy Skills (TILLS) | 6 months after initial evaluation
  It was developed by Nelson and his colleagues to assess the oral and written language skills of school-age children (6-18). The test consists of 15 subtests that measure different stages of oral and written language skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol Mega University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gernsbacher MA, Kaschak MP. Neuroimaging studies of language production and comprehension. Annu Rev Psychol. 2003;54:91-114. doi: 10.1146/annurev.psych.54.101601.145128. Epub 2002 Jun 10. PMID 12359916
- [Background] Safi D, Lefebvre P, Nader M. Literacy acquisition: Reading development. Handb Clin Neurol. 2020;173:185-199. doi: 10.1016/B978-0-444-64150-2.00017-4. PMID 32958173
- [Background] Habib S. Learning and Teaching British Values [Internet]. Cham: Springer International Publishing; 2018 [a.yer 15 Aralık 2023]. Erişim adresi: http://link.springer.com/10.1007/978-3-319-60381-0
- [Background] Dehaene S, Cohen L, Morais J, Kolinsky R. Illiterate to literate: behavioural and cerebral changes induced by reading acquisition. Nat Rev Neurosci. 2015 Apr;16(4):234-44. doi: 10.1038/nrn3924. Epub 2015 Mar 18. PMID 25783611
- [Background] Houde O, Rossi S, Lubin A, Joliot M. Mapping numerical processing, reading, and executive functions in the developing brain: an fMRI meta-analysis of 52 studies including 842 children. Dev Sci. 2010 Nov;13(6):876-85. doi: 10.1111/j.1467-7687.2009.00938.x. PMID 20977558
- [Background] Bernhardt EB. "Reading in the Foreign Language." Listening, Reading, and Writing: Analysis and Application. Barbara HW, editör. Northeast Conference on the Teaching of Foreign Languages; 1986. 93- 11 s.
- [Background] Just MA, Carpenter PA. A capacity theory of comprehension: individual differences in working memory. Psychol Rev. 1992 Jan;99(1):122-49. doi: 10.1037/0033-295x.99.1.122. PMID 1546114
- [Background] Whitehurst G, Lonigan C. Emergent literacy: Development from pre-readers to readers. Neuman S, Dickinson K, editörler. New York: Guilford: Handbook of early literacy research; 2001. 11-29 s.
- [Background] Nouwens S, Groen MA, Kleemans T, Verhoeven L. How executive functions contribute to reading comprehension. Br J Educ Psychol. 2021 Mar;91(1):169-192. doi: 10.1111/bjep.12355. Epub 2020 May 22. PMID 32441782
- [Background] Miller MR, Müller U, Giesbrecht GF, Carpendale JI, Kerns KA. The contribution of executive function and social understanding to preschoolers' letter and math skills. Cognitive Development. 2013;28(4):331-49.
- [Background] Gallen CL, Schaerlaeken S, Younger JW; Project iLEAD Consortium; Anguera JA, Gazzaley A. Contribution of sustained attention abilities to real-world academic skills in children. Sci Rep. 2023 Feb 15;13(1):2673. doi: 10.1038/s41598-023-29427-w. PMID 36792755
- [Background] McClelland MM, Acock AC, Piccinin A, Rhea SA, Stallings MC. Relations between Preschool Attention Span-Persistence and Age 25 Educational Outcomes. Early Child Res Q. 2013 Apr 1;28(2):314-324. doi: 10.1016/j.ecresq.2012.07.008. Epub 2012 Aug 3. PMID 23543916
- [Background] Hoover WA, Gough PB. The simple view of reading. Read Writ. 01 Haziran 1990;2(2):127-60.
- [Background] Daigle D, Armand F, Armand F, Armand F. L'approche bilingue et l'apprentissage de la lecture chez les sourds. Revue de l'Association canadienne de linguistique appliquée (ACLA). 2004;7(1):23-38.
- [Background] Perfetti C, Stafura J. Word Knowledge in a Theory of Reading Comprehension. Scientific Studies of Reading. 2014;(18):22-37.
- [Background] Raatz U, Mhling R. Frankfurter tests für Fünfjhrige-Konzentration (FTF-K). Weinheim Beltz. 1971 [a.yer 15 Aralık 2023]; Erişim adresi: https://www.scirp.org/reference/referencespapers?referenceid=1626613
- [Background] Kaymak S. Yuvaya giden beş yaşındaki çocuklarla dikkat toplama çalışmaları [Yayınlanmamış yüksek lisans tezi]. [Ankara]: Ankara Üniversitesi Sosyal Bilimler Enstitüsü; 1995.
- [Background] Kurt M, Karakaş S. Sağ serebral hemisferin bilişsel işlevlerine duyarlı üç nöropsikolojik testin özellikleri ve aralarındaki ilişkiler. 3P Dergisi. 2000;(8):251-65.
- [Background] Kılıç BG, Irak M, Koçkar Aİ, Şener S, Karakaş S. İşaretleme Testi Türk Formu'nun 6-11 Yaş Grubu Çocuklarda Standardizasyon Çalışması. Klinik Psikiyatri Dergisi. 2002;5(4):213-28.
- [Background] Kurt M. Sağ serebral hemisferin bilişsel işlevlerine duyarlı nöropsikolojik testlerin faktör yapısının incelenmesi [Yayınlanmamış yüksek lisans tezi]. [Ankara]: Hacettepe Üniversitesi; 1998.
- [Background] Lezak M. Neuropsychological Assessment. 3. Baskı. New York: Oxford University Press; 1995.
- [Background] Weintraub S, Mesulam MM. Right cerebral dominance in spatial attention. Further evidence based on ipsilateral neglect. Arch Neurol. 1987 Jun;44(6):621-5. doi: 10.1001/archneur.1987.00520180043014. PMID 3579679
- [Background] Wechsler D, The Wechsler Intelligence Scale for children. 3. bs. San Antonio, TX: The Psychological Corporation; 1991.
- [Background] Uluç S, Öktem F, Erden G, Gençöz T, Sezgin N. Wechsler Çocuklar için Zeka Ölçeği-IV: Klinik Bağlamda Zekanın Değerlendirilmesinde Türkiye için Yeni Bir Dönem. Türk Psikoloji Yazıları. 14(28):49-57.
- [Background] Cameron Ponitz CE, McClelland MM, Jewkes AM, Connor CM, Farris CL, Morrison FJ. Touch your toes! Developing a direct measure of behavioral regulation in early childhood. Early Childhood Research Quarterly. 01 Nisan 2008;23(2):141-58.
- [Background] McClelland MM, Cameron CE, Duncan R, Bowles RP, Acock AC, Miao A, Pratt ME. Predictors of early growth in academic achievement: the head-toes-knees-shoulders task. Front Psychol. 2014 Jun 17;5:599. doi: 10.3389/fpsyg.2014.00599. eCollection 2014. PMID 25071619
- [Background] Akyürek G, Bumin G. Turkish Adaptation of The Executive Functions and Occupational Routines Scale (EFORTS) and Its Validity And Reliability. Dev Med Child Neurol. 2017;(59):2-18.
- [Background] Harber JR. Perception and perceptual-motor integration: there is a difference. Percept Mot Skills. 1979 Dec;49(3):917-8. doi: 10.2466/pms.1979.49.3.917. PMID 530792
- [Background] Colarusso R, Hammil D. Motor-free perception test (MVPT-3). California: Academic Therapy Publication; 2003.
- [Background] Mailend ML, Plante E, Anderson MA, Applegate EB, Nelson NW. Reliability of the Test of Integrated Language and Literacy Skills (TILLS). Int J Lang Commun Disord. 2016 Jul;51(4):447-59. doi: 10.1111/1460-6984.12222. Epub 2016 Mar 27. PMID 27018642
- [Background] Metin Ş, Aral N. Motor beceriden bağımsız görsel algı testi-3: Geçerlik güvenirlik çalışması. Çankırı Karatekin Üniversitesi Sosyal Bilimler Enstitüsü Dergisi. 2012;4(2):57-72.
- [Background] Atavasun Uysal S. Az Gören Çocuklarda İki Farklı Görsel Algılama Tedavisinin Etkinliğinin Karşılaştırılması [Doktora Tezi]. [Ankara]: Hacettepe Üniversitesi; 2009.